CLINICAL TRIAL: NCT04392570
Title: The Effect of Ramadan Fasting on Serum Osmolarity in Patients With Type 2 Diabetes
Brief Title: The Effect of Fasting on Serum Osmolarity in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Mirac Vural Keskinler, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: RAMADAN2020
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Type2 Diabetes
Keywords: fasting, osmolarity, fluid loss
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fasting group: patients with type 2 diabetes who prefer to fast during Ramadan
  Interventions: Diagnostic Test: Fasting
- Non-fasting group: patients with type 2 diabetes who are otherwise healthy and have no contraindications for fasting but prefer not to fast

INTERVENTIONS:
Diagnostic Test: Fasting — blood samplings will be taken 08:00 am and again 2 hours before breaking the fast
  Groups: Fasting group

SUMMARY:
In Ramadan, Muslims perform a special kind of fasting. Their fasting start with the first lights of the sunrise and end with the sunset. Especially in summer, it is a real challenge, as the time for fasting might be as long as 18 hours, and hot weather might cause severe dehydration. This might be dangerous, especially in patients with diabetes. Serum osmolarity is a good surrogate marker to evaluate the body's fluid content. We aimed to investigate if summertime Ramadan fasting causes further fluid loss in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Till recently, it was assumed that patients with type 2 diabetes have to eat frequently, especially to avoid hypoglycemia, which is still true if they are using sulphonylurea or insulin. Especially because patients with diabetes often have one or more diabetic complications, they were advised against Ramadan fasting, as it is not allowed to eat or drink anything for long hours. There are increasing data supporting intermittent fasting, where individuals won't eat anything for 12-18 hours but are permitted to drink sugar-free beverages. The new antihypoglycemic agents have the advantage of causing very low or no hypoglycemia, which allows these patients to eat less frequently. There are studies about the metabolic effect of intermittent fasting in patients with type 2 diabetes, but we don't have enough data for the safety of religious fasting where no kind of fluid intake is allowed. In this study, we aimed to investigate the effect of fasting on the fluid status of diabetic patients. To this effect, we used serum osmolarity to determine fluid status. The patients who preferred to fast were our study group, and the patients who were healthy otherwise but preferred not to fast were our control group. In Ramadan, contrary to the customary practice of intermittent fasting, fasting starts with the sunrise and continues till sunset. We planned to take the first blood sample at 10 am and the second blood sample at 06 pm in both groups and compare the serum osmolarity accordingly.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes
* will accept to give two different blood samples
* will prefer to fast during Ramadan ( for the intervention group)
* will prefer not to fast during Ramadan ( for the control group)
* have good glycemic control

Exclusion Criteria:

* if the patients are not eligible for fasting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients who were attending to the clinics of diabetes in a medical faculty
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
To compare the serum osmolarities of patients with type 2 diabetes who are fasting for 17 hours and who are not fasting. | 1 month
  osmolarity is the measure of solute concentration. In our study we used it as a surrogate marker for fluid loss during fasting

CONTACTS AND LOCATIONS:
Overall Officials: Mirac Vural Keskinler, MD, Principal Investigator — IMU Doctoral program
Locations (1):
- IMU Goztepe Education and Research Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keskinler MV, Dincer B, Caklili OT, Oguz A. The effect of Ramadan fasting on serum osmolality in diabetic patients. J Pak Med Assoc. 2023 Apr;73(4):767-770. doi: 10.47391/JPMA.3517. PMID 37051980